CLINICAL TRIAL: NCT01582360
Title: Pharmacokinetics of Anti-infectives in Critically Ill Patients in Need of Continuous Renal Replacement Therapy (CRRT) or Without CRRT
Brief Title: 2012_PharmacoCRRT-study:Pharmacokinetics of Anti-infectives in Critically Ill Patients in Need of Continuous Renal Replacement Therapy (CRRT)
Acronym: PharmacoCRRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/10076; 2011/10076 (OUSH) (Other: 2011/10076 (Oslo University Hospital))
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Critically Ill; Acute Renal Failure; Acute Kidney Injury
Keywords: critical illness; pharmacokinetics; CRRT; CVVH; CVVHD; CVVHDF; antiinfectives; antibiotics; minimum inhibitory concentration; bacterial killing; pharmacodynamics; PK/PD index
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- antiinfectiva: vancomycin: 80 patients Completed.
- antiinfectiva: meropenem: 80 patients recruiting
- antiinfectiva: flukonazol: 80 patients
- antiinfectiva: cefotaxim: 80 patients
- antiinfectiva: benzylpenicilline: 80 patients
- antiinfectiva: tazobactam piperacillin: 80 patients recruiting
- antiinfectiva: cloxacillin: 80 patients
- antiinfectiva: ciprofloxacin: 80 patients

SUMMARY:
The main purpose of the study is to examine if changes in pharmacokinetics of important antiinfectives in Critically Ill patients in need of continuous renal replacement therapy (CRRT), causes inadequate concentrations in plasma.

The effect of different modus of CRRT: CVVH and CVVHD will be compared, as well as type of filter, filter lifetime etc.

Hypothesis: The risk of incorrect dosage of antiinfectives - to low/ to high- is increased in critically ill patients receiving CRRT. Inadequate plasma concentrations of antiinfectives may contribute to increased mortality in this group.

DETAILED DESCRIPTION:
The main purpose of the study is to examine if changes in pharmacokinetics of important antiinfectives in Critically Ill patients in need of continuous renal replacement therapy (CRRT), causes inadequate concentrations in plasma.

The effect of different modus of CRRT: CVVH and CVVHD will be compared, as well as type of filter, filter lifetime etc.

Hypothesis: The risk of incorrect dosage of antiinfectives - to low/ to high- is increased in critically ill patients receiving CRRT. Inadequate plasma concentrations of antiinfectives may contribute to increased mortality in this group.

The antiinfectives to be examined are meropenem, fluconazol, cefotaxim, ciprofloxacin, tazobactam-piperacillin, vancomycin,penicillin,cloxacillin.

Endpoints:

1. Measured plasma concentrations of antiinfectives are sufficient for maximal microbial killing.
2. To identify the most important variability factors for plasma concentrations of antiinfectives in patients receiving CRRT
3. Establish and validate a routine for measurement of vital antiinfectives.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to ICU in need of antiinfectives:

   1. in need of CRRT
   2. without acute kidney failure
2. requirement for antiinfectives> 72 hrs
3. Age > 18 yrs
4. signed informed consent

Exclusion Criteria:

1. Acute or chronic renal failure not in need of CRRT
2. Age < 18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to the ICU at Oslo University Hospital, in need of treatment with antiinfectives.
Sampling Method: Non-Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Sub-therapeutic levels of measured antiinfectiva | 72 hours
  Pharmacokinetic/pharmacodynamic index achieved for each antiinfectiva

SECONDARY OUTCOMES:
SOFA-score | 72 hrs
  Sequential organ failure assessment, first 3 days after initiation of therapy
Mortality | 90-days

CONTACTS AND LOCATIONS:
Overall Officials: Elin Helset, MD PhD, Study Chair — Oslo University Hospital; Jan Fr Bugge, MD PhD, Principal Investigator — Oslo University Hospital; Elizabeth von der Lippe, MD PhD, Principal Investigator — Oslo University Hospital; Hilde Ma Sporsem, cand pharm, Principal Investigator — Sykehusapotekene Oslo; Yvonne Lao, cand pharm, Principal Investigator — Sykehusapotekene Oslo
Locations (1):
- Oslo University Hospital, Oslo, Norway